CLINICAL TRIAL: NCT05831735
Title: Adapted Physical Activity as Complementary Treatment to Alleviate the Symptoms of Endometriosis? The CRESCENDO Program (inCRease Physical Exercise and Sport to Combat ENDOmetriosis)
Brief Title: The CRESCENDO Program (inCRease Physical Exercise and Sport to Combat ENDOmetriosis)
Acronym: CRESCENDO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Upper Alsace University (Other)
Collaborators: National Research Agency, France (Other); EndoFrance (independant association for endometriosis) (Unknown); Hôpital de la Croix-Rousse (Other); University Hospital, Strasbourg, France (Other); University Hospital, Grenoble (Other); Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Principal Investigator, Geraldine Escriva-Boulley, Principal investigator, Upper Alsace University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ANR-22-CE36-0002-01
Record Dates: First submitted 2023-02-03; First posted 2023-04-26 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Endometriosis; Quality of Life
Keywords: endometriosis,; physical activity,; education,; pain; videoconferencing
MeSH Terms: conditions — Endometriosis; Motor Activity; Pain | interventions — Exercise; Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): This group will be provided with a video showing the movement to do in case of pain, or endometriosis crisis
- Physical activity (Experimental): This group will be provided with a video showing the movement to do in case of pain, or endometriosis crisis + with 1h to 3 h of adapted physical activity delivered by videoconference.
  Interventions: Behavioral: Physical activity
- Physical activity and education (Experimental): This group will be provided with a video showing the movement to do in case of pain, or endometriosis crisis + with 1h to 3 h of adapted physical activity delivered by videoconference + 6 session of educational and discussion groups
  Interventions: Behavioral: Physical activity; Behavioral: Physical activity and education

INTERVENTIONS:
Behavioral: Physical activity — The 6-month APA program is supervised via the videoconference platform and/or carried out independently based on a personalized written program that is updated weekly. The program is based on structured sessions alternating 3 types of PA: aerobic sessions, stretching sessions and muscle strengthening sessions (to be practiced following the teacher's oral or written instructions).
  The sessions last from 20 minutes to 1 hour and are of low to moderate intensity depending on the initial level of fitness. The sessions are structured, adapted and progressive. During the sessions, the exercises are adapted according to the means and materials available to the patients at home or in their immediate environment.
  The patients will be progressively led to practice in an autonomous way (i.e., without supervision) but following an adapted, personalized and structured program. These PA sessions can be declared afterwards to the PA teacher,(duration and the exercises actually performed).
  Arms: Physical activity; Physical activity and education
Behavioral: Physical activity and education — In addition to the intervention in physical activity, the people participating in this program will benefit from 6 months of educational activity (EA). The EA program includes 6 sessions scheduled according to the patients' availability in groups and by videoconference.
  Following their entry into the study and their allocation to the programs (1 month maximum), the patients will be invited to a first individual EA session, in order to establish an educational diagnosis (1 hour). This session will allow for an assessment of their needs and the presentation of the workshops. Then, between the second and the sixth month following randomization, patients will benefit from 5 collective EA sessions per group of 6 patients maximum (1h30 to 2h). These sessions will be about PA, nutrition, pain management. An individual session will be held at the end of the intervention and will allow for an educational assessment.
  Arms: Physical activity and education

SUMMARY:
Symptoms due to endometriosis cause psychological distress and interpersonal difficulties. However, studies on the psychological and social consequences of endometriosis are scarce, none has investigated life-partners' view of the disease and its consequences, and all adopt cross-sectional designs.

Research highlights the beneficial effects of adapted physical activity (APA), on chronic diseases. Thus, APA may have a beneficial effect on the symptoms and the psychological and social consequences of endometriosis. However, studies questioning the link between PA and endometriosis are rare. The scarcity of studies can be explained by the fact that due to the painful symptoms caused by the disease; women avoid practicing. It is worth noticing that, in the specific context of endometriosis, the barriers and facilitators to PA are not clearly identified. Otherwise, due to their cross-sectional design, it is not possible for these studies to establish a causal link between PA and endometriosis. A RCT is needed to test the effects of PA on endometriosis and its consequences.

The investigators' ambition is to fill these gaps in the existing literature and to allow a more comprehensive view of the phenomena at play in the relation between PA and endometriosis. To this end, the investigators will seek to achieve 2 objectives:

1. to identify the perceived effects of the disease on different areas of patients' lives, specifically areas related to PA, and to examine the reasons why patients are or are not physically active using a mixed methodology. Life-partners and women who do not suffer from this disease will also be involved in this study.
2. to investigate the effects of an APA program which includes therapeutic patient education (TPE) on 3 primary outcomes: perceived pain, QoL, and PA. A complementary aim is to determine the effect of the program on psychosocial and motivational variables, and on physiological variables.

Patients will be randomly assigned to 3 groups: (1) control, (2) APA, (3) APA + TPE. The investigators hypothesize that the program could (H1) complement current treatments for endometriosis by reducing pain, increasing QoL, increasing PA, (H2) have beneficial effects on patients' physical, psychological and social health as well as physiological factors.

DETAILED DESCRIPTION:
a. Objectives and research hypothesis

1. Endometriosis and its consequences Endometriosis is a chronic disease characterized by growth of endometrial tissue outside the uterine cavity which affects 200 million women (The investigators use the word "women" generically. However, this study takes into account gender identity. In other words, a person with endometriosis may identify as a man, as woman or no/other gender.) worldwide. In addition to infertility, one of the most common symptoms of endometriosis is pelvic chronic pain. Evidence has suggested that these symptoms result from a local inflammatory peritoneal reaction caused by ectopic endometrial implants that undergo cyclic bleeding. This disease generates significant health care costs (e.g., 9,5 billion in France) because there is no definite cure for it and its management involves pain related treatment and/or surgery. Research showed that these treatments are only relatively effective in reducing pain.

   This pain can cause psychological distress and interpersonal difficulties that are as difficult to live with as the pain itself. Compared to women who do not suffer from endometriosis, women with this disease develop a lower sense of femininity, altered body image, higher levels of stress, depression and anxiety. These factors affect their quality of life (QoL) and can have deleterious effects on the response to treatment. Interpersonal relationships are also impacted such as romantic, professional and social relationships, because the symptoms make it difficult to move and carry out daily activities. However, studies on the psychological and social consequences of endometriosis are scarce, few have investigated life-partners' view of the disease and its consequences, and all adopt cross-sectional designs.
2. The effects of physical activity on endometriosis: a question for further investigation In their recent publication, INSERM (L'Institut national de la santé et de la recherche médicale) highlights the beneficial effects of regular physical activity (PA) and adapted physical activity (APA) on chronic diseases. Research suggested that (A)PA may have a beneficial effect on the physical symptoms and the psychological and social consequences of these diseases, thus may be also in endometriosis context. However, studies questioning the link between PA and endometriosis (and its symptoms) are rare, cross-sectional, and their results are inconsistent. The scarcity of studies can be explained by the fact that due to the painful symptoms caused by the disease; women do not practice much PA spontaneously and autonomously or even avoid practicing. In addition to this difficulty, widely recognized barriers to PA (i.e., lack of time, lack of adequate and nearby infrastructure, and low self-confidence and motivation for PA) can also contribute to the low level of PA. It is worth noticing that, in the specific context of endometriosis, the barriers and facilitators to the practice of PA are not clearly identified. Otherwise, due to their cross-sectional design, it was not possible for these studies to establish a causal link between PA and endometriosis. A randomized controlled trial (RCT) is needed to test the effects of (A)PA on the symptoms of endometriosis and its consequences.
3. Summary of scientific barriers to be lifted

Based on previous research and their limits, there are three major scientific barriers to be lifted regarding the investigation of the link between (A)PA and endometriosis:

1. There is a need to better understand the psychological and social factors associated to endometriosis. For instance, consequences of endometriosis on these factors and the impact of the disease in romantic relationships (i.e., on the patient and on her life partner2) need to be more documented. Some of these factors could be related to patient PA or could mediate or moderate the relation between endometriosis (and its symptoms) and PA.
2. Although barriers of PA are well known, in the context of endometriosis the barriers and facilitators to the practice of PA are not clearly identified. Given the specificity of this disease which only affect women and its impact on body functioning and body perception, this topic deserves to be investigated.
3. Otherwise, due to their scarcity and their cross-sectional design, it was not possible for previous studies to strongly establish a causal link between PA and, endometriosis and its symptoms. Conducting a RCT may help to overcome this limitation.

4. Objectives and hypotheses The investigators' ambition for this original work is to fill these gaps in the existing literature and to allow a more comprehensive view of the phenomena at play in the relation between PA and endometriosis. For this purpose, The investigators will use a multimethodological design and a multidisciplinary approach in one of the first intervention study led with patients who suffer from endometriosis.

Within two work packages (WP) the investigators will identify the perceived effects of the disease specifically those related to PA, and investigate the reasons why patients are or are not physically active using qualitative and quantitative methodologies (WP1). Otherwise, this first study will allow investigating and thus identifying the barriers and leverages to PA in the specific context of endometriosis.

This information could be particularly interesting in the development of the WP2. Indeed, in WP2 which is an exploratory study, The investigators will investigate the effects of an APA program delivered by videoconferencing which include therapeutic patient education (TPE) on PA and sedentary behaviors (SED), on perceived pain, QoL, and on patients' physical, physiological (inflammatory status and oxidative stress) social and psychological health.

The primary objectives of the WP2 were to investigate the effects of the CRESCENDO program on PA and SED but also on perceived pain and QoL. The investigators choose to also investigate pain and QoL as primary outcomes because their evolution are key elements in endometriosis setting. Thus, the primary outcomes were defined as the proportion of patients who

1. achieve the internationally recommended level of PA international recommendations, i.e., at least 150 minutes per week of moderate to vigorous PA
2. indicate a decrease in their perceived pain level (at least 1 point or 1 centimeter on visual analogue scale)
3. indicate an increase in their QoL level (at least 20 points)

The investigators hypothesize that the CRESCENDO program could (H1) complement current treatments for endometriosis by increasing PA and reducing SED, reducing pain (due to the decrease of inflammatory status), increasing QoL, (H2) have beneficial effects on patients' physical, psychological and social health as well as physiological factors. Finally, a program combining APA and TPE will be more effective than one that offers these interventions separately (H3). It is worth noticing that, the questionnaire which will be propose in WP2 will be similar to those proposed in WP1. The investigators expect to find coherent results, that is, The investigators expect to explain part of the WP2 results based on WP1 results.

In view of the expected benefits for the patients benefiting from the program, the investigators hope that the results of this study will lead to the generalization of the integration of APA and TPE programs into endometriosis care protocols. These practices could be considered as a complement, or even an alternative, to treatments to reduce healthcare costs. The use of videoconferencing to deliver APA programs would remove barriers to PA related to the availability and proximity of sports facilities and scheduling constraints, as much as allow the continuity of the practice even if the health context imposes a lockdown (e.g., COVID-19), while allowing for a group practice that is adapted and emotionally reassuring. Finally, the inclusion of chronic diseases among the diseases for which patient can benefit of a medical prescription for sport (i.e., APA) and the launch of the national strategy against endometriosis lead by C. Zacharopoulou in Marsh 2021, confirmed in January 2022, emphasized the importance of these related topics: endometriosis and APA. The investigators hope the results of this study to be informative to select the type of care which is the most adapted and efficient to endometriosis patients, that is to shed light on the importance of proposing a comprehensive care which could have an impact on physical and psychosocial variables.

ELIGIBILITY:
Inclusion Criteria:

* 18 years,
* sexually active,
* having endometriosis confirmed by laparoscopy or MRI (or saliva test if approved by health authorities),
* reporting moderate to significant functional difficulties and pain (between 4 and 10 / 10 points on visual analogue scale), and
* having free access to the internet to participate in the APA and TPE sessions, and fill in the questionnaires.

Exclusion Criteria:

* having a disabling disease other than endometriosis (cancer, fibromyalgia, arthritis, ...),
* a BMI higher than 35,
* not experiencing major difficulties related to the disease,
* having surgery or Medically Assisted Procreation scheduled within 9 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived pain and fatigue | before the start of the intervention and at the end of the intervention (6 months)
  10 point scale from 0 (none) to 10 (extreme pain or fatigue), today, last week en during an endometriosis episode
Change in Perceived Quality of life; Endometriosis Health Profile 30 | before the start of the intervention and at the end of the intervention(6 months)
  Likert scale questionnaire about quality of life in different life domains (1 to 7 )
Change in Physical activity (PA) ; International Physical Activity Questionnaire & International Sedentary Assessment Tool | before the start of the intervention and at the end of the intervention(6 months)
  complete the number of hour and minutes spend in Light, moderate and vigourous PA and in sedentary behaviors

SECONDARY OUTCOMES:
Change in self image | before the start of the intervention and at the end of the intervention(6 months)
  likert scale questionnaire about self perceptions (1 to 7 )
Change in perceived social support | before the start of the intervention and at the end of the intervention(6 months)
  Likert scale questionnaire about social support from family, friends, life partner (1 to 5 )
Change in stereotype | before the start of the intervention and at the end of the intervention(6 months)
  Likert scale questionnaire about the perception of the possibility for person with endometriosis to perform PA (1 to 7)
Change in motivation | before the start of the intervention and at the end of the intervention(6 months)
  likert scale questionnaire (1 to 7) self-determination theory (Bhavsar et al., 2020 ; Boiché et al. 2016), self efficacy (Everett et al., 2009)

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine Escriva, Phd, Principal Investigator — Upper Alsace University
Locations (1):
- Upper Alsace University, Mulhouse, Escriva-Boulley, France

IPD SHARING:
Plan to Share IPD: Yes
anonymisation
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The study protocol and the inform consent form will be shared at the beginning of the study (march 2023). The report will be avalaible at the end of the study (march 2024).
  The document will be available for 10 years.
Access Criteria: This information will be made avalable on open research websites (sport arxiv, psycarxiv, PCI movement...) and on request by email to the first authors or the principal investigator.

REFERENCES:
- [Derived] Escriva-Boulley G, Philip CA, Warembourg S, Lenotre L, Flore P, Faure P, Michy T, Letouzey V, Arnold C, Piluso C, Chalmel L, Kacem R, Blum GF, Detayrac R, Trocme C, Brigaud I, Herbach U, Branche P, Faller E, Chalabaev A. Effects of a physical activity and endometriosis-based education program delivered by videoconference on endometriosis symptoms: the CRESCENDO program (inCRease physical Exercise and Sport to Combat ENDOmetriosis) protocol study. Trials. 2023 Nov 27;24(1):759. doi: 10.1186/s13063-023-07792-1. PMID 38012776